CLINICAL TRIAL: NCT04987242
Title: An Inpatient, Placebo-Controlled Study of ALLN-346 (Engineered Urate Oxidase) in Hyperuricemic Subjects
Brief Title: An Inpatient Study of ALLN-346 (Engineered Urate Oxidase) in Hyperuricemic Subjects (Study 201)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-346-201
Record Dates: First submitted 2021-07-26; First posted 2021-08-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hyperuricemia; Gout; Chronic Kidney Diseases
MeSH Terms: conditions — Hyperuricemia; Gout; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Study population includes generally healthy subjects with hyperuricemia without CKD, and those with eGFR of mild-moderate CKD. The maximal tolerated dose from the MAD study in normal healthy volunteers (Study 102) will be administered. The study is comprised of two Parts. Under optional Part 2, only subjects with eGFR of CKD Stages 2- 3a.
Who Masked: Participant, Investigator
Masking Description: Subjects, Investigators and laboratories involved in the conduct of the study will be blinded to subject treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLN-346 (Engineered Urate Oxidase) (Experimental): ALLN-346 is novel urate oxidase provided as capsules for oral administration: 5 capsules thrice daily (TID) for a total of 15 capsules per day will be evaluated for 7 days
  Interventions: Drug: ALLN-346
- Placebo (Placebo Comparator): Matching placebo capsules for oral administration: 5 capsules thrice daily (TID) for a total of 15 capsules per day will be evaluated for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLN-346 — ALLN-346 (Engineered Urate Oxidase) is an orally administered, novel urate oxidase; provided as capsules for oral administration
  Other Names: Engineered urate oxidase
  Arms: ALLN-346 (Engineered Urate Oxidase)
Drug: Placebo — Matched placebo capsules are similar in weight and appearance to the ALLN-346 capsules
  Other Names: Matching placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this Phase IIa study is to evaluate the safety and tolerability of ALLN-346 in subjects with hyperuricemia in an inpatient, controlled setting.

DETAILED DESCRIPTION:
This is a Phase II, 7-day, randomized, double-blind, placebo-controlled study of orally administered ALLN-346 in subjects with hyperuricemia, with subpopulations to include generally healthy hyperuricemic subjects with normal kidney function and those with mild to moderate chronic kidney disease (CKD). Study will take place at a clinical pharmacology unit (CPU). The study will have two Parts. Part 1 will include subjects with serum urate ≥ 6.8 mg/dL and eGFR ≥ 60 mL/minute/1.73 m2 (subjects with eGFR of stage 2 CKD and with normal kidney function). Part 2 will include subjects with serum urate ≥ 6.8 mg/dL and eGFR 45-100 mL/minute/1.73 m2 (eGFR of CKD Stages 2- 3a).

The study will evaluate safety, tolerability, pharmacokinetics (lack of absorption) and pharmacodynamics of ALLN-346.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 55 years
* sUA level ≥ 6.8 mg/dL at Screening (hyperuricemia), with or without a diagnosis of gout
* Not pregnant, not capable of pregnancy, not nursing, and agrees to use an effective method of contraception; males subjects must agree to abstain from sperm donation
* Normal non-clinically significant abnormalities in vital signs
* Normal clinical laboratory test results and ECG, which are not considered to be clinically significant

Exclusion Criteria:

* Screening eGFR of <60 mL/minute/1.73 m2 for Part 1, and for Part 2 Screening eGFR outside the range of 45-100 mL/minute/1.73 m2.
* History or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, urological, or psychiatric disorders.
* Presence or history of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines
* Currently taking any urate-lowering medication within 4 weeks prior to Day 1 (first dosing day)
* Prior uricase therapy or exposure to recombinant uricase
* Clinically significant abnormal findings on electrocardiogram (ECG)
* Positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody
* Received treatment with or exposure to an Investigational drug or device within 30 days - prior to or during Screening
* Prior dosing in ALLN-346 clinical study
* Per Investigator judgment, is not an ideal clinical study candidate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 21 days per Study Part
  Number of of participants with treatment emergent adverse events

SECONDARY OUTCOMES:
Serum ALLN-346 | 8 days
  Serum concentration of ALLN-346 (ng/mL)

OTHER OUTCOMES:
Serum Urate | 8 days
  Serum urate [mg/dL]

CONTACTS AND LOCATIONS:
Overall Officials: C Tosone, MS, RAC, Study Director — Allena Pharmceuticals
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No